CLINICAL TRIAL: NCT03283787
Title: A Single Site Randomized, Clinical Trial Comparing the Concomitant Use of MicroMatrix® With Cytal™ Wound Matrix 2-Layer to Standard of Care in Patients With Stage 3 or 4 Pressure Injuries
Brief Title: Comparing Concomitant Use of ACell MicroMatrix® and ACell Cytal™ to Standard of Care in Stage 3 or 4 Pressure Injuries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Integra LifeSciences Corporation (Industry)
Collaborators: St Vincent's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA2016-001
Record Dates: First submitted 2017-09-13; First posted 2017-09-14 (Actual); Results first posted 2020-11-16 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-03

CONDITIONS: Pressure Ulcers Stage III; Pressure Ulcer, Stage IV; Pressure Ulcer
Keywords: Pressure Ulcer; ACell; ACell MicroMatrix®; ACell Cytal™; Extracellular Matrix; Urinary Bladder Matrix; Wound
MeSH Terms: conditions — Pressure Ulcer; Wounds and Injuries | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Group 1 (Active Comparator): MicroMatrix® and Cytal™ Wound Matrix 2-Layer
  Interventions: Device: MicroMatrix® and Cytal™ Wound Matrix 2-Layer
- Group 2 (Active Comparator): MicroMatrix® and Cytal™ Wound Matrix 2-Layer plus NPWT
  Interventions: Device: MicroMatrix® and Cytal™ Wound Matrix 2-Layer plus NPWT
- Group 3 (Active Comparator): Negative Pressure Wound Therapy
  Interventions: Device: Negative Pressure Wound Therapy

INTERVENTIONS:
Device: MicroMatrix® and Cytal™ Wound Matrix 2-Layer — MicroMatrix® and Cytal™ Wound Matrix 2-Layer
  Arms: Group 1
Device: MicroMatrix® and Cytal™ Wound Matrix 2-Layer plus NPWT — MicroMatrix® and Cytal™ Wound Matrix 2-Layer plus NPWT
  Arms: Group 2
Device: Negative Pressure Wound Therapy — Negative Pressure Wound Therapy
  Arms: Group 3

SUMMARY:
The purpose of this study is to evaluate incidence of complete epithelialization in stage 3 & 4 pressure ulcers using ACell products.

DETAILED DESCRIPTION:
A three arm, parallel-design, randomized study comparing 2 experimental arms to a single control arm. The primary comparison will be Group 1 (MicroMatrix® and ACell Cytal™ Wound Matrix 2-Layer vs. Group 3 (NPWT) to determine if Group 1 is superior to Group 3. NPWT is the standard of care (SOC) for patients with Stage 3 or 4 pressure ulcers and is the active control arm for the study.

A secondary comparison will be conducted comparing Group 2 (MicroMatrix® and ACell Cytal™ Wound Matrix 2-Layer plus NPWT) vs. Group 3 (NPWT) to determine if Group 2 is superior to Group 3.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form by subject or legally authorized representative.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Male or female patients that are ≥ 21 years of age.
4. Body Mass Index (BMI) <45.
5. At least one Stage 3 or 4 pressure injury (NPUAP Staging Guidelines) present at the Screening and/or Treatment Visit located in any of the following regions:

   1. Occipital
   2. Back
   3. Flank
   4. Upper Extremity

   i. Arm ii. Elbow iii. Wrist iv. Hand e. Sacral f. Hip g. Gluteal h. Ischial i. Lower Extremity i. Leg ii. Knee iii. Ankle iv. Heel v. Foot
6. Surface dimensions of pressure injury must be between 9 to 64 cm2 inclusive (as measured prior to treatment using a cm-scale ruler). The longest dimension must not exceed 10 cm; depth must not exceed 5 cm.
7. Wound must be >5 cm from the anus if colostomy not performed.
8. For lower extremity ulcers: Adequate arterial blood flow and perfusion near the site of the injury (the foot is warm to the touch and has palpable pulses), per Investigator judgement.
9. Confirmed pressure injury versus moisture-associated skin damage or friction injury.
10. Ability to maintain an intact occlusive dressing for 4-7 days with reinforcement without contamination of urine or stool.
11. Confirmed fecal (Colostomy) and/or urine incontinence (Foley) maintenance/management, if necessary.
12. Consent to off-loading (turns) from pressure sites a minimum of every 2 hours (if possible).
13. Consent to sharp debridement of necrotic tissue in the wound bed unless the wound has already undergone debridement within 5 days prior to the Treatment Visit.
14. For females of reproductive potential (defined as females ≤ 55 years of age): Negative pregnancy test required prior to surgical debridement per hospital procedures.

Exclusion Criteria:

1. Surgical treatment of pressure injury 30 days prior to the Treatment Visit and/or pressure injury in previously irradiated areas.
2. Inability to manage fecal and/or urine incontinence or patient refusal of its maintenance/management (as determined medically necessary). Patient may be rescreened and enrolled if urinary and/or fecal continence status or management change after failure to comply with requirement.
3. Allergy or hypersensitivity to materials in porcine-based study products (per subject report) or personal preference.
4. Currently treated for an active malignant disease.
5. Prior diagnosis of active malignant disease, and is less than 1 year disease-free.
6. History of malignancy within the wound.
7. Presence of any conditions that are contraindicated with NPWT.
8. Any condition associated with a wound healing abnormality (e.g.: connective tissue disorder or immune disorder).
9. Dermatologic comorbid disease (e.g., cutis laxa or collagen vascular disease).
10. Bleeding diathesis.
11. Patients with primary treatment ulcers from burns (from exposure to high heat) or venous leg ulcers. A patient may have concomitant non-pressure ulcers present in non-pressure ulcer treatment regions.
12. Received biological-based therapy in any pressure wound within 3 months of the Treatment Visit.
13. Severe or significant hypoalbuminemia (albumin <2.5 g/dL, and/or pre-albumin <5 mg/dL), or hypoproteinemia (protein <6 g/dL).
14. Moderate to severe anemia (Hgb <7 g/dL).
15. Severely uncontrolled diabetes mellitus (defined as HA1C >12%).
16. Subject report of concurrent participation in another clinical trial that involves an investigational drug or device that would interfere with this study.
17. Subject report of previous participation in other interventional wound healing clinical investigation within 60 days prior to the Screening Visit.
18. The subject has any physical or psychiatric condition that in the Investigator's opinion would warrant exclusion from the study or prevent the subject from completing the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-09-25 (Actual); Study Completion 2019-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol Bowen-Wells, MD, Principal Investigator — Saint Vincent's Medical Center Riverside
Locations (1):
- Saint Vincent's Medical Center, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data

RESULTS

PARTICIPANT FLOW:
Groups:
- MicroMatrix® and Cytal™ Wound Matrix 2-Layer: Treatment protocol per PI SOC discretion utilizing study devices.
- MicroMatrix® and Cytal™ Wound Matrix 2-Layer Plus NPWT: Treatment protocol per PI SOC discretion utilizing study device plus NPWT.
- Negative Pressure Wound Therapy: Treatment protocol per PI SOC discretion.
Period: Overall Study
Arm/Group | MicroMatrix® and Cytal™ Wound Matrix 2-Layer | MicroMatrix® and Cytal™ Wound Matrix 2-Layer Plus NPWT | Negative Pressure Wound Therapy
Started | 20 | 20 | 20
Completed | 17 | 13 | 13
Not Completed | 3 | 7 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Total
Number analyzed (Participants) | 20 | 20 | 20 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 9 | 5 | 25
  >=65 years | 9 | 11 | 15 | 35
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 10 | 21
  Male | 14 | 15 | 10 | 39
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 13 | 9 | 10 | 32
  White | 7 | 11 | 9 | 27
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Complete Epithelialization
Description: Number of participant wounds with complete epithelialization by 12 weeks. Complete wound closure (epithelialization) determination based on PI assessment.
Time Frame: 12 weeks
Measure: Number; unit: No of wounds w/ complete epithelization
Groups:
- MicroMatrix® and Cytal™ Wound Matrix 2-Layer; MicroMatrix® and Cytal™ Wound Matrix 2-Layer Plus NPWT; Negative Pressure Wound Therapyroup 3: Treatment protocol per PI discretion
Arm/Group | MicroMatrix® and Cytal™ Wound Matrix 2-Layer | MicroMatrix® and Cytal™ Wound Matrix 2-Layer Plus NPWT | Negative Pressure Wound Therapyroup 3
Number analyzed (Participants) | 20 | 20 | 20
No of wounds w/ complete epithelization | 2 | 1 | 0

2. Secondary Outcome: Time to Complete Wound Epithelization
Description: Time to complete wound epithelization between groups.
Time Frame: 12 weeks
Population: The secondary outcome analysis was confounded due to the heterogeneity of the data and amplified by the small samples size. The study data heterogeneity resulted from the clinically distinct wounds and subject risk profiles that limited interpretability and utility. This challenge was validated by an independent third party review.
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Rate of Wound Epithelization
Description: Rate of wound epithelization between groups
Time Frame: 12 weeks
Population: as for outcome 2
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 Months
Arm/Group | Group 1 | Group 2 | Group 3
All-Cause Mortality (participants affected / at risk) | 0/20 | 2/20 | 4/20
Serious Adverse Events (participants affected / at risk) | 2/20 | 2/20 | 5/20
Other Adverse Events (participants affected / at risk) | 9/20 | 18/20 | 19/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=20) | Group 2 (N=20) | Group 3 (N=20)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Blunt Trauma (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hip/Femur Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Seizure (General disorders) | 0 (0) | 0 (0) | 1 (1)
Complications related to pneumonia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral Arterial Disease and End stage renal disease (General disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=20) | Group 2 (N=20) | Group 3 (N=20)
Bleeding (General disorders) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 5 (5) | 9 (20) | 12 (25)
Periwound Maceration (Skin and subcutaneous tissue disorders) | 5 (6) | 15 (27) | 19 (52)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Wound Recurrence (General disorders) | 0 (0) | 1 (1) | 0 (0)
Wound contamination, secondary to diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Wound Vac Leaking (General disorders) | 0 (0) | 0 (0) | 1 (1)
Lethargic (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoglycemia and AMS (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-08): https://cdn.clinicaltrials.gov/large-docs/87/NCT03283787/Prot_SAP_000.pdf